CLINICAL TRIAL: NCT05001347
Title: A Phase 2 Clinical Study of TJ004309 in Combination With Atezolizumab (TECENTRIQ®) in Patients With Advanced or Metastatic Ovarian Cancers and Selected Advanced Solid Tumors
Brief Title: A Clinical Study of TJ004309 With Atezolizumab (TECENTRIQ®) in Patients With Ovarian Cancer and Selected Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: I-Mab Biopharma US Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJ004309STM103
Record Dates: First submitted 2021-07-12; First posted 2021-08-11 (Actual); Results first posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Ovarian Cancer; Head and Neck Cancer; Non Small Cell Lung Cancer; Gastrointestinal Cancer; Triple Negative Breast Cancer; Ovarian Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms; Head and Neck Neoplasms; Carcinoma, Non-Small-Cell Lung; Gastrointestinal Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TJ004309 and Atezolizumab (Experimental): TJ004309 20 mg/kg Q3W in combination with atezolizumab 1200 mg Q3W
  Interventions: Drug: TJ004309

INTERVENTIONS:
Drug: TJ004309 — Antibody to CD73

SUMMARY:
This is a multicenter, open label, Phase 2 study of TJ004309 in combination with atezolizumab in patients with advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
This is a multicenter, open label, Phase 2 study of TJ004309 in combination with atezolizumab in patients with advanced or metastatic solid tumors. This clinical study includes two cohorts: Cohort 1 will include Immuno-Oncology (IO) treatment naïve ovarian cancer (OC) patients who have progressed on or after platinum therapy; and Cohort 2 will include patients with head and neck squamous cell carcinoma (HNSCC), non-small cell lung cancer (NSCLC), gastrointestinal cancer (GC), triple negative breast cancer (TNBC), or ovarian carcinoma (OC) with PD-L1 expression ≥ 1%. Additional cohorts for selected tumor types might be added later.

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1: Patients with histologically confirmed epithelial ovarian cancer, fallopian tube, or primary peritoneal cancer subjects with any high-grade serous component, progressed on or after platinum-containing therapy and not eligible for further platinum containing treatment (platinum-resistant, platinum-refractory disease defined by progression of disease on a platinum-containing regimen or recurrence of disease within 180 days of receiving the last dose of platinum-based treatment).
* Cohort 2: Patients with selected tumor types that have relapsed or progressed after 2 lines of therapy or who are ineligible for other standard of care (SOC) therapies:

  1. Histologically or cytologically confirmed metastatic NSCLC
  2. Histologically or cytologically confirmed recurrent or metastatic HNSCC (oral cavity, oropharynx, hypopharynx, or larynx)
  3. Histologically or cytologically confirmed metastatic or non-resectable advanced metastatic gastric or gastroesophageal adenocarcinoma
  4. Histologically or cytologically confirmed unresectable, locally advanced or metastatic TNBC (confirmed HER2-negative, estrogen receptor-negative and progesterone receptor-negative)
  5. Histologically confirmed ovarian cancer of all high-grade epithelial types who are IO treatment naïve and have progressed after 3 months on or after platinum-containing therapy
  6. PD-L1 expression Tumor Proportion Score (TPS) ≥ 1% for NSCLC and Combined Proportion Score (CPS) ≥ 1% for all other tumor types
  7. A 28-day washout period after the completion of programmed death-1 (PD-1)/PD-L1 therapy
  8. Patients should have no more than 5 prior lines of therapies
* Cohort 2 - (Optional for the ovarian cohort) Pre-treatment fresh tumor biopsies and paired treatment fresh tumor biopsies will be collected from at least 5 patients. Biopsy must be excisional, incisional, or core.

Exclusion Criteria:

* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g. cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], OX 40 [Tumor necrosis factor receptor superfamily, member 4 (TNFRSF4)], CD137 [tumor necrosis factor receptor superfamily member 9 (TNFRSF9)]) (only applies to ovarian cancer patients in Cohorts 1 and 2)
* Disease progression within 3 months of starting anti-PD-1 and anti-PD-L1 inhibitors
* Known active or chronic Hepatitis B or Hepatitis C, other hepatitides (non-alcohol steatohepatitis, alcohol or drug-related, autoimmune) serology at screening or cirrhosis
* Active autoimmune disease requiring systemic treatment within the past 12 months
* Active interstitial lung disease (ILD) or pneumonitis or a history of ILD
* Brain involvement with cancer, spinal cord compression, carcinomatous meningitis, or new evidence of brain or leptomeningeal disease; unless the lesion(s) have been radiated or resected, are considered fully treated and inactive, are asymptomatic, and no steroids have been administered for CNS disease over the 7 days prior to study treatment
* Angina, myocardial infarction (MI), symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack TIA), arterial embolism, pulmonary embolism, percutaneous transluminal coronary angioplasty (PTCA), or coronary artery bypass grafting (CABG) within 6 months prior to study treatment
* Known human immunodeficiency virus (HIV) unless CD4+ T cell count > 350 cells/μL with an undetectable viral load

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2023-02-08 (Actual); Study Completion 2023-02-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Arizona Oncology Associates, Tucson, Arizona
  - Innovative Clinical Research Institute, Whittier, California
  - Medical Oncology Hematology Consultants, PA, Newark, Delaware
  - Illinois Cancer Specialists, Arlington Heights, Illinois
  - Women's Cancer Care, Covington, Louisiana
  - Maryland Oncology Hematology, Rockville, Maryland
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Duke Cancer Center, Durham, North Carolina
  - Tri County Hematology and Oncology Associates, Massillon, Ohio
  - Texas Oncology - Arlington North, Arlington, Texas
  - Texas Oncology - Austin Central, Austin, Texas
  - Texas Oncology - Forth Worth Cancer Center, Fort Worth, Texas
  - Texas Oncology - The Woodlands, Gynecologic Oncology, The Woodlands, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Northwest Cancer Specialists, Vancouver, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Platinum resistant or refractory IO naive ovarian carcinoma (OC)
  TJ004309 20mg/kg Q3W and atezolizumab 1200 mg/flat dose Q3W
- Cohort 2: HNSCC, NSCLC, GC, TNBC, OC
  TJ004309 20 mg/kg Q3W and atezolizumab 1200 mg/flat dose Q3W
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 17 | 8
Completed | 3 | 2
Not Completed | 14 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 17 | 8 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 6 | 14
  >=65 years | 9 | 2 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (10.84) | 60.0 (11.35) | 63.2 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 3 | 20
  Male | 0 | 5 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 16 | 6 | 22
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 13 | 6 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants] — United States
  participants
    United States | 17 | 8 | 25

OUTCOME MEASURES:

1. Primary Outcome: To Assess the Efficacy of TJ004309 Combined With Atezolizumab in a Cohort of Patients With Platinum-resistant IO Naive Ovarian Carcinoma and a Separate Biomarker Enriched Cohort of Subjects With Selected Tumor Types
Description: Anti-tumor activity of the combination of TJ004309 and atezolizumab was measured by objective response rate (ORR) based on RECIST 1.1
Time Frame: Up to 66 weeks
Population: Efficacy evaluable analysis set was defined as all patients who received at least one dose of study drug and undergo at least one post-baseline tumor assessment. Patients who died before the first scheduled post-baseline tumor assessment were also included in the efficacy evaluable analysis set- only 23 of the 25 subjects were efficacy evaluable per this definition.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 15 | 8
Participants | 1 | 0

2. Secondary Outcome: o Assess the Efficacy of TJ004309 Combined With Atezolizumab in a Cohort of Patients With Platinum-resistant IO Naive Ovarian Carcinoma and a Separate Biomarker Enriched Cohort of Subjects With Selected Tumor Types
Description: Anti-tumor activity of the combination of TJ004309 and atezolizumab was measured by objective response rate (ORR) based on iRECIST.
Time Frame: Up to 66 weeks
Population: Overall number of participants is the number of subjects who had at least one response assessment (iRECIST) from N=6 out 15 in Cohort 1 and N=4 out of 8 in Cohort 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 6 | 4
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 15 months
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 4/17 | 2/8
Serious Adverse Events (participants affected / at risk) | 7/17 | 4/8
Other Adverse Events (participants affected / at risk) | 0/17 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=17) | Cohort 2 (N=8)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 1
Infusion-related reaction (Injury, poisoning and procedural complications) | 0 | 1
Cardiac Failure congestive (Cardiac disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Biliary Obstruction (Hepatobiliary disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/47/NCT05001347/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-22): https://cdn.clinicaltrials.gov/large-docs/47/NCT05001347/SAP_001.pdf